CLINICAL TRIAL: NCT02643316
Title: Morning-Only 4 Liter Polyethylene Glycol vs. Split Dose for Afternoon Colonoscopies, a Randomized Endoscopist-Blinded Prospective Study
Brief Title: Morning-Only 4 L PEG vs Split Dose Prep for Afternoon Colonoscopies, Endoscopist-Blinded Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Fernando Castro, Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FLA 15-092
Record Dates: First submitted 2015-12-29; First posted 2015-12-31 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Same day 4 L preparation of PEG (Active Comparator): Receive 1 gallon (4 L) of Polyethylene Glycol (PEG) preparation on the morning of the colonoscopy.
  Interventions: Drug: Same day 4 L preparation (Polyethylene Glycol)
- Split dose 4 L preparation of of the PEG (Active Comparator): Receive the split-dose regimen. Will take half (2 L) of the PEG preparation the evening before colonoscopy and half (2 L) of the PEG preparation on the morning of the procedure.
  Interventions: Drug: Split dose 4 L preparation (Polyethylene Glycol)

INTERVENTIONS:
Drug: Same day 4 L preparation (Polyethylene Glycol) — Receive 1 gallon (4 L) of Polyethylene Glycol preparation on the morning of the colonoscopy.
  Other Names: PEG bowel prep
  Arms: Same day 4 L preparation of PEG
Drug: Split dose 4 L preparation (Polyethylene Glycol) — Receive the split-dose regimen. Will take half (2 L) the preparation the evening before colonoscopy and half (2 L) on the morning of the procedure.
  Other Names: PEG bowel prep
  Arms: Split dose 4 L preparation of of the PEG

SUMMARY:
Comparison of quality of preparation of colonoscopy in patients taking same day 4L preparation vs. 4 L split dose preparation in patients scheduled for an afternoon colonoscopy procedure.

DETAILED DESCRIPTION:
The aim of colorectal cancer screening is to reduce mortality. This can be effectively achieved by colonoscopy with direct visualization of the entire colon to detect preneoplastic lesions such as adenomatous polyps. Bowel preparation quality is critical for the accuracy of colonoscopy, time required to complete the procedure and its success. On the other hand, poor quality of bowel preparation was shown to be associated with a lower adenoma detection rate. Prior studies have shown that time of colonoscopy is one of the major factors influencing bowel preparation quality with the afternoon colonoscopies being notable for a high failure rate. This failure rate is related to poor bowel preparation quality. Given that, the number of afternoon colonoscopies performed is still high due to the increased need for colonoscopies. Therefore, it is suggested that improving the bowel preparation quality can reduce failure rate of afternoon colonoscopies. Several studies on split-dose bowel preparation have shown that it is superior to the conventional day-before regimen, in terms of preparation quality and patient's tolerability. Another study on split-dose bowel preparation also showed that it is associated with a better adenoma detection rate, better polyp detection rate and colonoscopy completion rate. There also have been few studies comparing same day dose vs. day-before for afternoon colonoscopies and showed that same day was superior to day before.There is no data comparing quality of preparation of colonoscopy in patients taking same day 4L preparation vs. 4 L split-dose preparation for an afternoon colonoscopy.

Using a 4L PEG-ELS solution, the investigators aim to evaluate the efficacy and patient's tolerability for the same day versus split-dose regimen.

ELIGIBILITY:
Inclusion Criteria:

1. All patients above 18 years of age undergoing elective outpatient colonoscopy at CCF Florida who are scheduled for an afternoon colonoscopy procedure. All patients must have been prescribed a 4 L PEG based bowel preparation.

Exclusion Criteria:

1. Patients who had prior Colectomy or colon resection surgery.
2. Patients with confirmed diagnosis of impaired GI motility.
3. Chronic nausea or vomiting.
4. Severe constipation (=/<1 bowel movement per week).
5. Pregnancy.
6. Breast feeding.
7. Patients taking drugs which are known to influence GI motility.
8. Hospital inpatients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Quality of preparation (Ottawa score) | During the colonoscopy
  The quality of bowel preparation will be assessed for the 2 groups at the time of the colonoscopy using the Ottawa score for quality of preparation.

SECONDARY OUTCOMES:
Patient satisfaction with the bowel preparation (questionnaire). | Before the colonoscopy procedure.
  Patient satisfaction with the bowel preparation in the 2 groups will be assessed using an approved questionnaire at the time of pre-operative assessment of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Castro, M.D., Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castro FJ, Al-Khairi B, Singh H, Mohameden M, Tandon K, Lopez R. Randomized Controlled Trial: Split-dose and Same-day Large Volume Bowel Preparation for Afternoon Colonoscopy Have Similar Quality of Preparation. J Clin Gastroenterol. 2019 Nov/Dec;53(10):724-730. doi: 10.1097/MCG.0000000000001213. PMID 31021890